CLINICAL TRIAL: NCT03654599
Title: Effects of Digital Stories Intervention on Psychosocial Well-being for Cancer Patients and Caregivers Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Effects of Digital Stories Intervention on Psychosocial Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Mayo Clinic (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GR11968; R15CA213035 (NIH); NCT03440775 (obsolete NCT alias)
Record Dates: First submitted 2018-08-27; First posted 2018-08-31 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Bone Marrow Transplant; Information Disclosure; Hematopoietic Stem Cell Transplantation; Psychosocial Health; Depression; Anxiety; Stress; Narrative
Keywords: Digital Storytelling; Narrative; Cancer patients; Psychosocial health; bone marrow transplant
MeSH Terms: conditions — Depression; Anxiety Disorders; Narration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline and Digital Stories (DS) for patients (Experimental): In-person baseline surveys using the web-based data collection platform, Research Electronic Data Capture before the random assignment to DS arm. Eight Digital Stories Intervention (4 patient and 4 caregiver stories about hematopoietic stem cell transplantation (HCT) over the course of 4 weeks (2 videos per week) with a weekly email notification and reminder phone call. Each story was made with voice, images, and sound (3-5 minutes each).
  Interventions: Behavioral: Baseline Surveys; Behavioral: Digital Stories Intervention
- Baseline and Information Control (IC) for patients (Active Comparator): In-person baseline surveys using the web-based data collection platform, Research Electronic Data Capture (REDCap) before the random assignment to IC arm. Eight Information Control Intervention videos containing only information about post-HCT care (as opposed to story/narrative) over the course of 4 weeks (2 videos per week) with a weekly email notification and reminder phone call.
  Interventions: Behavioral: Baseline Surveys; Behavioral: Information Control Intervention
- Baseline and Digital Stories (DS) for caregivers (Experimental): In-person baseline surveys using the web-based data collection platform, Research Electronic Data Capture before the random assignment to DS arm. Eight Digital Stories Intervention (4 patient and 4 caregiver stories about hematopoietic stem cell transplantation (HCT) over the course of 4 weeks (2 videos per week) with a weekly email notification and reminder phone call. Each story was made with voice, images, and sound (3-5 minutes each).
  Interventions: Behavioral: Baseline Surveys; Behavioral: Digital Stories Intervention
- Baseline and Information Control (IC) for caregivers (Active Comparator): In-person baseline surveys using the web-based data collection platform, Research Electronic Data Capture (REDCap) before the random assignment to IC arm. Eight Information Control Intervention videos containing only information about post-HCT care (as opposed to story/narrative) over the course of 4 weeks (2 videos per week) with a weekly email notification and reminder phone call.
  Interventions: Behavioral: Baseline Surveys; Behavioral: Information Control Intervention

INTERVENTIONS:
Behavioral: Baseline Surveys — Baseline surveys contained a series of scaled questions, including sociodemographic variables (age, sex, cancer type, and etc), profile of mood states, social well-being, emotional processing and acceptance.
  Other Names: Baseline questionnaire
Behavioral: Digital Stories Intervention — Digital Stories Intervention Videos contain the following content: caregiver burden, positive and cognitive coping, support from other family and friends, fear of losing the patient, spirituality, guilt of being sick, and expressing emotions/feelings
  Other Names: Digital Storytelling; Narrative-based storytelling
  Arms: Baseline and Digital Stories (DS) for caregivers; Baseline and Digital Stories (DS) for patients
Behavioral: Information Control Intervention — Information Control Intervention Videos include Information about post-HCT. The topics in the IC include specific guidelines to return to wellness post HCT through (1) an exercise plan, (2) a nutrition (dietary) plan, (3) pain management, (4) information about the complications, (5) caregiver responsibilities, (6) social support, (7) preventing from infections, and (8) symptom management. Participants randomized to the IC will receive the full set of DS modules only after the final 3-month post-intervention data collection point has passed and they can view them as desired.
  Arms: Baseline and Information Control (IC) for caregivers; Baseline and Information Control (IC) for patients

SUMMARY:
Patients and caregivers undergoing hematopoietic stem cell transplantation often continue to experience anxiety, depression, isolation, and other psychosocial distress. A narrative-based digital stories intervention has shown promise in a pilot study with breast cancer patients in helping to alleviate emotional distress. This study is designed to test digital stories to be viewed and discussed by other HCT patients/caregivers as a psychosocial intervention in a randomized controlled trial and to test the effects of digital stories on how 110 patient and caregiver dyads (N=220) undergoing one of the most rigorous and aggressive treatments cope with treatment-related distress through supportive open dyadic communication and emotional expression.

DETAILED DESCRIPTION:
Patients and caregivers undergoing hematopoietic stem cell transplantation (HCT) are at particular risk for reduced psychological and social well-being due to the rigorous and unique nature of the transplant experience, such as prolonged immunosuppression and multiple post HCT complications resulting in frequent hospitalizations. However, few studies have evaluated interventions to alleviate psychosocial distress for both patients and caregivers, and those have yielded inconclusive results. A narrative-based (storytelling) approach may be an effective intervention tool for HCT patients and caregivers coping with psychosocial distress. The preliminary data show that stories shared by individuals in which a range of emotional expression or resolutions are described, may have beneficial effects on emotional well-being. In a recent pilot study of a 3-day digital storytelling workshop, investigators produced a series of digital videos with narratives from a panel of post-HCT patients. The purpose of this study is to use these digital stories (DS), to be viewed and discussed by HCT patient/caregiver dyads, as a therapeutic intervention and to examine influences on both patients' and caregivers' psychosocial status. This cost-effective, non-invasive, and easy-to-deliver psychosocial support vehicle has never been formally tested as an intervention for HCT patients or patient-caregiver dyads.

To build upon investigators' preliminary studies and to pilot test the efficacy of this series of DS, 110 adult patients undergoing HCT at the Mayo Clinic Arizona and patient respective adult caregivers (N=220 total participants) will be randomized to either (a) an intervention using DS (dyadic exposure to four 5-minute modules) or (b) an information control (IC) video group (dyadic exposure to four videos containing only information about post-HCT care) followed by encouragement to discuss as a dyad. Exposure will occur once per week over 4 weeks via a secure web-based data collection platform (REDcap) with a weekly email notification and reminder phone call. Using investigator's model of Narrative Effects on Socio-Emotional Well-Being, we will also examine expected mediating factors to determine how stories may "work" to reduce psychosocial distress by fostering emotional processing, acceptance, and dyadic disclosure of emotions.

ELIGIBILITY:
Patient Inclusion Criteria:

* age 18 or older
* recently underwent Hematopoietic cell transplantation (HCT) (within a month after hospital discharge)
* must be able to speak, read, and write in English
* access to a working phone and e-mail account

Patient Exclusion Criteria:

* no primary caregiver
* cognitive impairment that prohibits completion of study assessment
* visual or hearing impairment
* other (e.g., provider non-approval or logistical constraints such as patient moving out of town)

Caregiver Inclusion Criteria:

* age 18 or older
* family caregivers who are identified as a primary caregiver by a patient
* have primary responsibility for the care of patients throughout the HCT process
* Must be able to speak, read, and write in English
* Access to a working phone and e-mail account

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Kim, Ph.D, Principal Investigator — Arizona State University
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four enrolled participants were excluded from the study before assignment to groups due to patients' health issues (e.g., readmitted to the hospital, illness, and/or complications after the transplant).
Groups:
- Baseline and Digital Stories (DS): In-person baseline surveys using the web-based data collection platform, Research Electronic Data Capture before the random assignment to DS arm. Eight Digital Stories Intervention (4 patient and 4 caregiver stories about hematopoietic stem cell transplantation (HCT) over the course of 4 weeks (2 videos per week) with a weekly email notification and reminder phone call. Each story was made with voice, images, and sound (3-5 minutes each).
  Baseline Surveys: Baseline surveys contained a series of scaled questions, including sociodemographic variables (age, sex, cancer type, and etc), profile of mood states, social well-being, emotional processing and acceptance.
  Digital Stories Intervention: Digital Stories Intervention Videos contain the following content: caregiver burden, positive and cognitive coping, support from other family and friends, fear of losing the patient, spirituality, guilt of being sick, and expressing emotions/feelings
- Baseline and Information Control (IC): In-person baseline surveys using the web-based data collection platform, Research Electronic Data Capture (REDCap) before the random assignment to IC arm. Eight Information Control Intervention videos containing only information about post-HCT care (as opposed to story/narrative) over the course of 4 weeks (2 videos per week) with a weekly email notification and reminder phone call.
  Baseline Surveys: Baseline surveys contained a series of scaled questions, including sociodemographic variables (age, sex, cancer type, and etc), profile of mood states, social well-being, emotional processing and acceptance.
  Information Control Intervention: Information Control Intervention Videos include Information about post-HCT. The topics in the IC include specific guidelines to return to wellness post HCT through (1) an exercise plan, (2) a nutrition (dietary) plan, (3) pain management, (4) information about the complications, (5) caregiver responsibilities, (6) social support, (7) preventing from infections, and (8) symptom management. Participants randomized to the IC will receive the full set of DS modules only after the final 3-month post-intervention data collection point has passed and they can view them as desired.
Period: Overall Study
Arm/Group | Baseline and Digital Stories (DS) | Baseline and Information Control (IC)
Started (The Enrollment number includes all participants (both patients and caregivers). 106 participants = 53 patient-caregiver dyads.) | 106 | 92 (92 individuals = 46 patient/caregiver dyads)
Completed | 78 | 70
Not Completed | 28 | 22
Not completed — Lost to Follow-up | 14 | 12
Not completed — Death | 8 | 6
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Baseline and Information Control (IC) for Patients; Baseline and Information Control (IC) for Caregivers: n-person baseline surveys using the web-based data collection platform, Research Electronic Data Capture (REDCap) before the random assignment to IC arm. Eight Information Control Intervention videos containing only information about post-HCT care (as opposed to story/narrative) over the course of 4 weeks (2 videos per week) with a weekly email notification and reminder phone call.
  Baseline Surveys: Baseline surveys contained a series of scaled questions, including sociodemographic variables (age, sex, cancer type, and etc), profile of mood states, social well-being, emotional processing and acceptance.
  Information Control Intervention: Information Control Intervention Videos include Information about post-HCT. The topics in the IC include specific guidelines to return to wellness post HCT through (1) an exercise plan, (2) a nutrition (dietary) plan, (3) pain management, (4) information about the complications, (5) caregiver responsibilities, (6) social support, (7) preventing from infections, and (8) symptom management. Participants randomized to the IC will receive the full set of DS modules only after the final 3-month post-intervention data collection point has passed and they can view them as desired.
- Total: Total of all reporting groups
Arm/Group | Baseline and Digital Stories (DS) for Patients | Baseline and Digital Stories (DS) for Caregivers | Baseline and Information Control (IC) for Patients | Baseline and Information Control (IC) for Caregivers | Total
Number analyzed (Participants) | 53 | 53 | 46 | 46 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual.
  years | 56.8 (14.3) | 56.4 (12.9) | 53.1 (14.2) | 51.4 (16.4) | 54.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual.
  Participants
    Female | 22 | 42 | 18 | 30 | 112
    Male | 31 | 11 | 28 | 16 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual.
  Participants
    Hispanic or Latino | 5 | 7 | 8 | 8 | 28
    Not Hispanic or Latino | 46 | 44 | 37 | 37 | 164
    Unknown or Not Reported | 2 | 2 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual.
  Participants
    American Indian or Alaska Native | 2 | 2 | 3 | 3 | 10
    Asian | 0 | 0 | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 2 | 2 | 1 | 1 | 6
    White | 46 | 46 | 38 | 37 | 167
    More than one race | 3 | 3 | 4 | 4 | 14
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual.
  Participants
    United States | 53 | 53 | 46 | 46 | 198
Education [Count of Participants; unit: Participants] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual.
  Participants
    High School | 4 | 6 | 13 | 9 | 32
    Some college | 20 | 18 | 15 | 18 | 71
    4-year college degree | 18 | 21 | 10 | 10 | 59
    Graduate degree | 11 | 8 | 8 | 9 | 36
Marital Status [Count of Participants; unit: Participants] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual.
  Participants
    Married | 39 | 39 | 34 | 31 | 143
    Never Married | 3 | 3 | 2 | 6 | 14
    Divorced, widowed or separated | 8 | 6 | 6 | 3 | 23
    Not married | 3 | 5 | 4 | 6 | 18
Employment Status [Count of Participants; unit: Participants] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual.
  Participants
    Employed full time | 25 | 21 | 17 | 16 | 79
    Employed part time | 2 | 7 | 2 | 7 | 18
    Not employed | 26 | 25 | 27 | 23 | 101
Health insurance [Count of Participants; unit: Participants] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual.
  Participants
    Private Coverage | 34 | 36 | 31 | 29 | 130
    Medicaid | 1 | 1 | 2 | 2 | 6
    Medicare | 16 | 15 | 7 | 14 | 52
    Other | 2 | 1 | 6 | 1 | 10
Cancer diagnosis [Count of Participants; unit: Participants] — Population: This baseline characteristic was only collected for patients
  Participants
    Multiple Myeloma: number analyzed (Participants) | 53 | 0 | 46 | 0 | 99
    Multiple Myeloma | 19 | 0 | 9 | 0 | 28
    Lymphoma: number analyzed (Participants) | 53 | 0 | 46 | 0 | 99
    Lymphoma | 10 | 0 | 10 | 0 | 20
    Myelodysplastic Syndrome: number analyzed (Participants) | 53 | 0 | 46 | 0 | 99
    Myelodysplastic Syndrome | 11 | 0 | 11 | 0 | 22
    Leukemia: number analyzed (Participants) | 53 | 0 | 46 | 0 | 99
    Leukemia | 10 | 0 | 14 | 0 | 24
    Other: number analyzed (Participants) | 53 | 0 | 46 | 0 | 99
    Other | 3 | 0 | 2 | 0 | 5
Transplant type [Count of Participants; unit: Participants]
  Autologous | 14 | 14 | 11 | 11 | 50
  Allogeneic | 39 | 39 | 33 | 33 | 144
Main source of support [Count of Participants; unit: Participants] — This baseline measure was assessed in both patients and caregivers. The unit of analysis is individual. Participants can select all that apply.
  Participants
    Spouse | 35 | 32 | 29 | 25 | 121
    Sibling | 8 | 2 | 9 | 1 | 20
    Son/Daughter | 22 | 4 | 13 | 7 | 46
    Friends | 9 | 2 | 7 | 3 | 21
    Parents | 10 | 9 | 9 | 6 | 34
    Other | 6 | 4 | 4 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline Profile of Mood States (POMS) Short Version (Emotional Well-being or /Reduction of Emotional Distress) at 4 Weeks
Description: Emotional Well-Being (Reduction of Emotional Distress) will be measured using the Profile of Mood States (POMS) short version (15 items, 5-point Likert scale; 0=not at all, 4=extremely). The POMS is one of the most frequently used and validated scales in studies of psychosocial interventions for cancer patients. The POMS Total Mood Disturbance (TMD) score has been shown to be most sensitive to interventions designed to facilitate emotional expression.The POMS consists of the TMD dimensions (tension-anxiety; depression-dejection; anger-hostility; and confusion-bewilderment) (Cronbach's a = .93) to be used in the current study as the primary outcome measure; and two others (fatigue-inertia; vigor-activity) will be documented. Total of Mood Disturbance= (anxious+depression+anger+fatigue)- vigor (Range from 12 to 48). The higher values represent a worse emotional well-being.
Time Frame: Baseline (T1), T2 (after 4-week intervention)
Population: HCT patients and caregivers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline and Digital Stories (DS) | Baseline and Information Control (IC)
Number analyzed (Participants) | 78 | 70
score on a scale
  Baseline | 3.3 (3.0) | 3.4 (3.2)
  Post-Intervention | 2.4 (3.1) | 2.8 (3.1)

2. Secondary Outcome: Changes From Baseline Emotional Well-being (Using the Emotional Acceptance Scale) at 4 Weeks
Description: The 13-item Emotional Acceptance (EA) Scale assesses the extent to which subjects are accepting toward their feelings, with statements such as "I naturally and easily attend to my feelings." Respondents estimate the percentage of time each statement is true, in increments of 10 (0 = never/not at all to 100 = always/perfectly; total score = mean item rating). In Dr. Weihs' sample of 91 breast cancer patients, internal consistency was strong (= .92), as was 15-month test re-test reliability (r = .58).
Time Frame: Baseline (T1), T2 (after 4-week intervention)
Population: HCT patients and caregivers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline and Digital Stories (DS) | Baseline and Information Control (IC)
Number analyzed (Participants) | 78 | 70
score on a scale
  Baseline | 2.8 (0.57) | 2.8 (0.59)
  Post-intervention | 3.1 (0.64) | 3.0 (0.49)

ADVERSE EVENTS:
Time Frame: At 1 month, 3 months
Description: Participants have been withdrawn because the patient died during the intervention period. Given this study was the dyad study, caregivers were also withdrawn when their patients passed. Due to this reason, results in the adverse event for each arm/group were combined.
Arm/Group | Baseline and Digital Stories (DS) for Patients | Baseline and Digital Stories (DS) for Caregivers | Baseline and Information Control (IC) for Patients | Baseline and Information Control (IC) for Caregivers
All-Cause Mortality (participants affected / at risk) | 4/53 | 4/53 | 3/46 | 3/46
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03654599/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03654599/SAP_001.pdf
  • Informed Consent Form (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT03654599/ICF_002.pdf